CLINICAL TRIAL: NCT01866787
Title: Baroreceptor Function and Inflammation in Relation to Orthostatic Intolerance During Early Mobilization After Elective Hip Arthroplasty
Brief Title: Study on Baroreceptor Function in Relation to Orthostatic Blood Pressure Regulation After Hip Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Oeivind Jans, M.D., Research Fellow, Rigshospitalet, Denmark
Other Study IDs: RH-4074-OJ3
Record Dates: First submitted 2013-02-04; First posted 2013-05-31 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Hypotension, Orthostatic; Total Hip Replacement
Keywords: Postoperative orthostatic intolerance; Surgical inflammatory response
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for Hemoglobin measurement and plasma for inflammatory markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort

SUMMARY:
The purpose of this observational study is to evaluate the baroreceptor function in relation to surgical inflammation and orthostatic intolerance after elective hip arthroplasty.

The main hypothesis is that baroreceptor function is attenuated after surgery and related to surgical inflammation.

DETAILED DESCRIPTION:
Orthostatic intolerance and hypotension is prevalent during early mobilization after major surgery.

This observational study aims to evaluate the baroreceptor function during using a standardized evaluation protocol before, 6- and 24 hours after elective primary unilateral hip-arthroplasty.

The study hypothesis is that baroreceptor function as expressed by the valsalva ratio is attenuated after surgery and related to surgical inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral hip arthroplasty
* 18 years or older
* Able to give informed consent

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class 3 or higher
* Chronic arrythmia (Atrial fibrillation or other arrythmia)
* Incompensated ischaemic heart disease
* Mobilization restriction due to surgical reasons
* Medical complications during admission requiring transferral to other department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective unilateral hip arthroplasty at Frederiksberg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in baroreceptor function from preoperatively to 6 hours after surgery | 6 hours after surgery
  Change in baroreceptor function as expressed by change in the blood pressure valsalva ratio during a standardized assessment before and 6 hours after surgery.

SECONDARY OUTCOMES:
Orthostatic response in blood pressure | Preoperative, 6 and 24 hours after surgery
  The response in systolic and diastolic blood pressure during postural change from supine to standing
Orthostatic response in heart rate variability | preoperative, 6 and 24 hours postoperative
  Heart rate variability during supine rest, sitting and standing as assessed by Spectral analysis.
Orthostatic intolerance | preoperative, 6 and 24 hours after surgery
  Orthostatic intolerance defined as the inability to sit or stand for 3 minutes due to presyncopal symptoms (Dizziness, Nausea, Blurred vision).
Inflammatory markers | preoperative, 6 and 24 hours postoperative
  Inflammatory markers (CRP and interleukin-6) measured at 3 separate timepoint: preoperative, 6- and 24 h after surgery
Orthostatic Hypotension | Preoperative, 6 and 24 hours postoperative.
  orthostatic hypotension defined according to international guidelines.
Baroreceptor function | On the day of surgery: preoperatively, 6- and 24 hours after surgery
  baroreceptor function as expressed by change in the blood pressure valsalva ratio during a standardized assessment

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Jans, M.D, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Frederiksberg Hospital, Department of orthopaedic surgery, Frederiksberg, Denmark